CLINICAL TRIAL: NCT03491735
Title: Patterns of Glaucoma in Glaucoma Subspecialty Clinics in Egypt and India in the Year 2018
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Collaborators: Sadguru Netra Chikitsalaya, Post Graduate Institute Of Ophthalmology (New SNC) (Other)
Responsible Party: Principal Investigator, Rana H. Amin, Assistant Lecturer of Ophthalmology, Kasr El Aini Hospital
Other Study IDs: 12CM
Record Dates: First submitted 2018-04-02; First posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Determining Patterns of Glaucoma in Glaucoma Sub-specialty Clinics in Two Countries: Egypt and India
Keywords: patterns; glaucoma; egypt; india; 2018
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Patients referred to glaucoma sub-specialty clinics in Kasr Al-Aini Hospital, Cairo University, Egypt in the year 2018
  Interventions: Other: collection of data from patient files
- Group B: Patients referred to glaucoma sub-specialty clinics in Sadguru Netra Chikitsalaya Postgraduate Institute of Ophthalmology, Mumbai, India in the year 2018
  Interventions: Other: collection of data from patient files

INTERVENTIONS:
Other: collection of data from patient files — recording of patient data and its input into an excel sheet from which statistics will be derived

SUMMARY:
In this study, we are aiming to identify the patterns of glaucoma observed and treated at Glaucoma Subspecialty Clinics of Kasr Al-Aini Hospital, Cairo University in Cairo, Egypt and corresponding clinics in Sadguru Netra Chikitsalaya Post Graduate Institute of Ophthalmology in Mumbai, Maharashtra, India during the year 2018. We are hoping that this study would provide an update on current statistics available on Indian population as well as provide novel numbers on the prevalence of glaucoma and its patterns in one of the largest tertiary care hospitals in Egypt. These results will then be compared to patterns observed in other epidemiological studies done in other countries.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to glaucoma sub-specialty clinics in the year 2018 in two centres: Kasr Al-Aini Hospital in Cairo and Sadguru Netra Chikitsalaya Postgraduate Institute of Ophthalmology in India

Exclusion Criteria:

* Patients younger than 18 years old.
* Patients with incomplete examination data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred to and following up in the glaucoma sub-specialty clinics in the year 2018 in two centres: Kasr Al-Aini Hospital in Cairo and Sadguru Netra Chikitsalaya Postgraduate Institute of Ophthalmology in India
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Patterns of Glaucoma | 12 months starting january 1st, 2018 til December 31st, 2018
  Determining patterns of glaucoma seen in one year in glaucoma sub-specialty clinics in two countries: Egypt and India
Demographic data | 12 months starting january 1st, 2018 til December 31st, 2018
  Determining demographic data with respect to age and gender in different types of glaucoma in each country

SECONDARY OUTCOMES:
Anti-glaucoma treatment | 12 months starting january 1st, 2018 til December 31st, 2018
  Determining details of anti-glaucoma treatment used in each country
Positive family history | 12 months starting january 1st, 2018 til December 31st, 2018
  Determining percentage of patients with positive family history in each country
Management decisions | 12 months starting january 1st, 2018 til December 31st, 2018
  Determining different management decisions taken by doctors in each country

CONTACTS AND LOCATIONS:
Locations (2):
- Kasr Al-Aini Hospital, Cairo University, Cairo, Egypt
- two centres: Kasr Al-Aini Hospital in Cairo and Sadguru Netra Chikitsalaya Postgraduate Institute of Ophthalmology, Mumbai, India

IPD SHARING:
Plan to Share IPD: Yes
statistics obtained from data collected
Supporting Information: Study Protocol, SAP
Time Frame: january 1st 2018 til december 31st 2018